CLINICAL TRIAL: NCT04696926
Title: Five-year Outcomes of Rapid-deployment Aortic Valve Replacement With the Edwards Intuity TM Valve: a Single-center Prospective Study
Brief Title: Five-year Outcomes of Rapid-deployment Aortic Valve Replacement With the Edwards Intuity TM Valve
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: CIL 2019-48
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Severe Aortic Valve Disease
Keywords: severe aortic stenosis; severe aortic regurgitation
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis; Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients who underwent an aortic valve replacement
  Interventions: Other: Edwards Intuity TM Valve implantation

INTERVENTIONS:
Other: Edwards Intuity TM Valve implantation — aortic valve replacement with an Edwards Intuity TM bioprosthesis

SUMMARY:
Objectives:

This report presents 5-year outcomes of the rapid-deployment Edwards Intuity TM valve in a single-center prospective study.

Methods:

All consecutive patients who underwent an aortic valve replacement with an Edwards Intuity TM bioprosthesis at La Timone Hospital, Marseille, France, were prospectively included between July 2012 and June 2015 and were followed for 5 years. The primary outcome was overall mortality at 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients implanted by the Intuity TM bioprosthesis
* For severe aortic valve stenosis or severe aortic regurgitation
* Including reoperation and combined surgery
* Between July 2012 and June 2015

Exclusion Criteria:

* absence of patient's authorization for anonymous publication of their clinical data for research purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 170 consecutive patients who underwent an aortic valve replacement with an Edwards Intuity TM bioprosthesis at La Timone Hospital, Marseille, France, were prospectively included between July 2012 and June 2015 and were followed for 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
5-year overall mortality | 5 years
  overall mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France